CLINICAL TRIAL: NCT04871867
Title: Assessement of Cardiac and Lung Consequences of COVID-19 Infection in the Professional Soccer Players: A Prospective Observational Study
Brief Title: Cardiac and Lung Assessment of Professional Soccer Players Following COVID-19 Disease
Status: Completed | Type: Observational
Sponsor: American Hospital of Paris (Other)
Responsible Party: Principal Investigator, Gilles BOCCARA, principal investigator, American Hospital of Paris
Other Study IDs: americanHparis
Record Dates: First submitted 2021-05-01; First posted 2021-05-04 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Covid19
Keywords: COVID19; athletes; cardiac assessment; lung CT-scanner; COVID19 cardiopulmonary consequences
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During this world COVID-19 outbreak, and according to the experience of team doctors, after their return, some players could have been affected by the SARS-cov2. Also, this study aims to clearly determine the condition of athletes at the end of lockdown after this COVID-19 crisis and the cardiorespiratory consequences in particular in those who have been affected by COVID-19 and the prevalence of acute myocarditis. The investigators assess in this observational study the cardiac and lung consequences of COVID-19..

DETAILED DESCRIPTION:
The global health crisis caused by the COVID-19 virus, beginning in November 2019, initially in China, has being marked by a rapid spread, numerous severe respiratory cases and an elevated mortality rate. Although that 85% on average of patients with SARS-cov2 are not symptomatic or poor symptoms, these people were not systematically tested by PCR and spontaneously recovered. However, at the end of lockdown, the challenge for the medical staff in each first league soccer team involves to assess their clinical health conditions including clinical evaluation, COVID-19 tests, chest CT, and cardiac function in order to detect potential anomalies. Especially, physicians should be cautious about the risk of acute viral myocarditis, often asymptomatic, in patients having COVID-19 with any or poor symptoms, reported in 7 to 28%. The risk could be a myocardial dysfunction, arrhythmic complications and/or sudden death during return to exercice.

In this observational study, the investigators included the soccer player after the spring lockdown. After firstly an exhaustive interview to assess the lockdown quality of the athlete, clinical status and potential mild or poor symptoms of COVID-19 during the outbreak, and secondly COVID-19 serology and regular PCR tests.

The athletes having a positive nasopharyngeal SARS-cov2 PCR and/or positive COVID-19 serology test, with or without symptoms, were included in the study. Up to 10 days after first positive PCR, a cardiac evaluation is done including EKG, cardiac ultrasound echography and stress test in running ground and Chest Computer Tomography (chest-CT). According to the results of cardiac tests and Lung CT-scan, these athletes also require Cardiac MRI to eliminate the risk of acute myocarditis.

ELIGIBILITY:
Inclusion Criteria:

* Professional soccer player
* age over 18 years

Exclusion Criteria:

* recent muscle injury (< 1 month)
* recent orthopedic surgery (< 3 months)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Since 2020 spring and during this COVID-19 outbreak, the Professional soccer player were assessed about the COVID-19 infection using the clinical tests, swab PCR Test and SARS-Cov2 serology. The athletes having COVID-19 infection were included in cardiac and lung evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Cardiac abnormalities | up to ten days following COVID-19 infection
  qualitative
acute myocarditis occurence | up to ten days following COVID-19 infection
  qualitative
COVID19 lung lesions | up to ten days following COVID-19 infection
  qualitative

SECONDARY OUTCOMES:
global occurrence of COVID19 | one year since march 2020
  qualitative

CONTACTS AND LOCATIONS:
Overall Officials: Gilles BOCCARA, MD, PhD, Principal Investigator — Sport and Health unit of American Hospital of Paris
Locations (1):
- American Hospital of Paris, Neuilly-sur-Seine, France

REFERENCES:
- [Background] Fang Y, Zhang H, Xie J, Lin M, Ying L, Pang P, Ji W. Sensitivity of Chest CT for COVID-19: Comparison to RT-PCR. Radiology. 2020 Aug;296(2):E115-E117. doi: 10.1148/radiol.2020200432. Epub 2020 Feb 19. No abstract available. PMID 32073353
- [Background] Toresdahl BG, Asif IM. Coronavirus Disease 2019 (COVID-19): Considerations for the Competitive Athlete. Sports Health. 2020 May/Jun;12(3):221-224. doi: 10.1177/1941738120918876. Epub 2020 Apr 6. No abstract available. PMID 32250193
- [Background] Eirale C, Bisciotti G, Corsini A, Baudot C, Saillant G, Chalabi H. Medical recommendations for home-confined footballers' training during the COVID-19 pandemic: from evidence to practical application. Biol Sport. 2020 Jun;37(2):203-207. doi: 10.5114/biolsport.2020.94348. Epub 2020 Apr 10. PMID 32508388
- [Background] Schellhorn P, Klingel K, Burgstahler C. Return to sports after COVID-19 infection. Eur Heart J. 2020 Dec 7;41(46):4382-4384. doi: 10.1093/eurheartj/ehaa448. No abstract available. PMID 32432700
- [Background] Kochi AN, Tagliari AP, Forleo GB, Fassini GM, Tondo C. Cardiac and arrhythmic complications in patients with COVID-19. J Cardiovasc Electrophysiol. 2020 May;31(5):1003-1008. doi: 10.1111/jce.14479. Epub 2020 Apr 13. PMID 32270559
- [Background] Siripanthong B, Nazarian S, Muser D, Deo R, Santangeli P, Khanji MY, Cooper LT Jr, Chahal CAA. Recognizing COVID-19-related myocarditis: The possible pathophysiology and proposed guideline for diagnosis and management. Heart Rhythm. 2020 Sep;17(9):1463-1471. doi: 10.1016/j.hrthm.2020.05.001. Epub 2020 May 5. PMID 32387246
- [Background] Kim JH. Screening Athletes for Myocarditis With Cardiac Magnetic Resonance Imaging After COVID-19 Infection-Lessons From an English Philosopher. JAMA Cardiol. 2021 Aug 1;6(8):950-951. doi: 10.1001/jamacardio.2020.7463. No abstract available. PMID 33443538
- [Background] Martinez MW, Tucker AM, Bloom OJ, Green G, DiFiori JP, Solomon G, Phelan D, Kim JH, Meeuwisse W, Sills AK, Rowe D, Bogoch II, Smith PT, Baggish AL, Putukian M, Engel DJ. Prevalence of Inflammatory Heart Disease Among Professional Athletes With Prior COVID-19 Infection Who Received Systematic Return-to-Play Cardiac Screening. JAMA Cardiol. 2021 Jul 1;6(7):745-752. doi: 10.1001/jamacardio.2021.0565. PMID 33662103